CLINICAL TRIAL: NCT05985915
Title: A Randomized, Double-blind 2-arm NEPTUNUS Extension Study to Assess the Long-term Safety and Efficacy of Ianalumab in Patients With Sjogrens Syndrome.
Acronym: NEPTUNUS-Ext
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736A2301E1; 2022-502966-26-01 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Sjogrens Syndrome
Keywords: Sjogrens Syndrome; ianalumab; VAY736; NEPTUNUS
MeSH Terms: conditions — Sjogren's Syndrome | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ianalumab Monthly (Experimental): Ianalumab 300 mg s.c. monthly
  Interventions: Drug: Ianalumab (VAY736)
- Ianalumab 3 Monthly (Experimental): Ianalumab 300 mg s.c. every three months and placebo once monthly between doses
  Interventions: Drug: Ianalumab (VAY736); Other: Placebo

INTERVENTIONS:
Drug: Ianalumab (VAY736) — Ianalumab 300 mg / 2 mL, PFS or AI, monthly or every 3 months, solution for injection for subcutaneous use
  Other Names: VAY736
Other: Placebo — Placebo 0 mg/2 mL PFS or AI, once monthly between doses of Ianalumab 3 monthly , solution for injection for subcutaneous Use
  Arms: Ianalumab 3 Monthly

SUMMARY:
The purpose of this study is to measure the long-term safety and tolerability of ianalumab in participants with Sjogrens syndrome who have previously completed treatment from one of two NEPTUNUS 1 year core studies (CVAY736A2301 [NCT05350072] or CVAY736A2302 [NCT05349214]).

* The study treatment is ianalumab 300 mg in a 2 mL pre-filled syringe (PFS) or in a 2 mL autoinjector (AI) for injection. All participants will receive ianalumab either monthly or every 3 months.
* The treatment duration will be 3 years with an additional up to 2-year safety follow-up. The total duration of this extension study will be up to 5 years.
* The visit frequency will be monthly during both the treatment period and mandatory follow-up, and then less frequently during the subsequent conditional follow-up.

Treatment of interest: The randomized treatment (ianalumab) will be received monthly or every 3 months. Participants assigned to treatment every 3 months will receive placebo every month between the ianalumab doses to maintain blinding.

Number of Participants: Approximately 600 participants from the NEPTUNUS core studies will be rolled over into the extension study.

Treatment Groups:There will be no screening period in this trial. From Week 48 of the NEPTUNUS core study, participants will be given the opportunity to consent to this extension study. From Week 52 of the NEPTUNUS core studies (i.e., Day 1 in the extension study), eligible participants will be assigned to either one of the treatment regimens:

* ianalumab 300 mg monthly or
* ianalumab 300 mg once every 3 months

Participants receiving placebo in either of the NEPTUNUS core studies will be randomized 1:1 to receive ianalumab 300 mg monthly or every 3 months starting from Week 60 and participants receiving ianalumab in either of the NEPTUNUS core studies will continue the same treatment in the extension study.

Ianalumab will be given as a subcutaneous injection from a 2 mL pre-filled syringe or a 2 mL autoinjector. Participants will be given the opportunity to self-inject at home on some visits after receiving training.

DETAILED DESCRIPTION:
The primary purpose of this 3-year treatment extension study is the continued evaluation of the safety and tolerability of treatment with ianalumab 300 mg monthly or every 3 months. An additional purpose is to explore the long-term efficacy of both dosing regimens of ianalumab 300 mg.

Trial Design: This is a multicenter, randomized, double-blind, phase 3 study to assess the long-term safety and tolerability of four treatment regimens of ianalumab in participants with Sjogrens syndrome who have taken part in and completed one of two NEPTUNUS core studies, NEPTUNUS-1 (CVAY736A2301) or NEPTUNUS-2 (CVAY736A2302). There will be no screening period in this trial. From week 48 of the NEPTUNUS core study, participants will be given the opportunity to consent to this extension study. Eligible participants will continue their assigned treatment to receive ianalumab 300 mg either monthly or every 3 months for up to 3 additional years of treatment beyond the 1-year core study period. After the treatment period, all participants will enter a follow-up period to be monitored for at least 20 weeks and then a conditional (if B-cell recovery criteria have not been met) follow-up period. The total post treatment follow-up period is up to 2 years.

Study Population: Participants with Sjogrens syndrome who have completed treatment in one of two NEPTUNUS core studies.

Study treatment assignment method: Participants randomized to ianalumab 300 mg monthly or every 3 months in one of the NEPTUNUS core studies will continue their assigned treatment. Participants randomized to placebo in the NEPTUNUS core studies will be randomized in a 1:1 ratio to either ianalumab 300 mg monthly or every 3 months.

Participants randomized to ianalumab 300 mg every 3 months will receive placebo (a dummy treatment) once monthly between doses.

Committees: An independent Data Monitoring Committee (DMC) will be utilized for safety review throughout the study. A steering committee will be formed to ensure overview of the study conduct.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to participation in the extension study.
2. Participants must have participated in either one of the two NEPTUNUS core studies, CVAY736A2301 or CVAY736A2302, and must have completed the entire treatment up to Week 48 without treatment discontinuation in core NEPTUNUS studies.
3. In the judgement of the Investigator, participants must be expected to clinically benefit from continued ianalumab therapy.

Exclusion Criteria:

1. Use of therapies excluded by the NEPTUNUS-1 and NEPTUNUS-2 study protocols (see NEPTUNUS studies protocols exclusion criteria in Section 5.2 for details).
2. Plans for administration of live vaccines during the study period.
3. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human Chorionic Gonadotropin (hCG) laboratory test.
4. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment during dosing and for 6 months after stopping of investigational drug. Highly effective contraception methods include:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   * Female bilateral tubal ligation, female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or total hysterectomy at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant.
   * Use of oral (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.

   In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

   Contraception should be used in accordance with locally approved prescribing information of concomitant medications administered.

   Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age-appropriate history of vasomotor symptoms). Women are considered of not child-bearing potential if they are post-menopausal or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child-bearing potential.

   If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the informed consent form (ICF).
5. United States (and other countries, if male contraception is locally required): Sexually active males, unless they agree to use barrier protection during intercourse with a woman of child-bearing potential, while taking study treatment. As condom use alone has a reported failure rate exceeding 1% per year, it is recommended that female partners of male study participants use a second method of birth control. Although ianalumab is not teratogenic and/or genotoxic, and not transferred to semen, male contraception is required, as requested by FDA.

Globally, for all sexually active males, contraception should be used in accordance with the locally approved prescribing information of concomitant medications administered.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2028-08-21 (Estimated); Study Completion 2030-07-18 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment-emergent AEs (TEAEs)/SAEs | Week 52 to Week 304
  Assessment of safety and tolerability of ianalumab (VAY736) in patients with active Sjogrens syndrome

SECONDARY OUTCOMES:
ESSDAI change from baseline | Over time up to Week 204
  EULAR Sjogren's syndrome disease activity index (ESSDAI) is a validated clinical disease outcome measure for Sjogrens that will be used in the study The instrument contains 12 organ-specific domains contributing to assessment of disease activity. For each domain, features of disease activity are scored by a clinician in 3 or 4 (Level 0=No disease activity to Level 3= high disease activity) levels according to their severity. These scores are then summed across the 12 domains in a weighted manner to provide the total score. The maximum possible score is 123.To calculate ESSDAI, all 12 organ domains must be individually assessed by a trained assessor (study Investigator) at every scheduled timepoint. This is to evaluate the long-term efficacy of VAY736 300 mg administered monthly or every 3 months.
Percentage of participants achieving ESSPRI ≤ 3 AND ≥ 1.5 points reduction from baseline | Over time up to Week 204
  The EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) questionnaire consists of three items to be given an activity level score between 0-10: pain (joint and/or muscle pain), fatigue and dryness (0 = no symptom at all and 10 = worst symptom imaginable
  ESSPRI is an established disease outcome measure for Sjogrens. It consists of three domains of dryness, pain and fatigue. The participant will assess severity of symptoms they experience on a single 0-10 numerical scale for each of the three domains. The ESSPRI score is defined as a mean of scores from the three scales: (dryness + pain + fatigue) /3.
Percentage of participants achieving meaningful improvement in the SSSD score | Over time up to Week 204
  The Sjogrens Syndrome Symptom Diary (SSSD) questionnaire consists of five (six for females) questions about symptoms of Sjögren's syndrome, each question given a score of 0-10 (0=no symptoms, 10=worst possible symptoms) where patient choose the one response that best describes how severe the symptom was at its worst in the PAST 24 HOURS. It includes six symptom items (eye dryness, mouth dryness, skin dryness, physical fatigue, muscle and/or joint pain, genital dryness), and applies a recall period of 24 hrs. The aim of the SSSD is to establish patient reported endpoints for the treatment of Sjogrens syndrome. Participants will complete the diary daily for 7 days prior to the scheduled dosing.
Pre-dose Ianalumab serum concentrations | pre-dose at Week 48 (from core study) and Week 64
  To show comparability of ianalumab Ctrough between 2x 1 mL PFS (from the NEPTUNUS core studies) and 1x 2 mL PFS for participants on continuous monthly treatment.
On-treatment Ianalumab serum concentrations | During treatment (from Week 52 to Week 204) and follow-up (From Week 208 to Week 304)
  To further assess the pharmacokinetics of ianalumab.
B-cell count measurement | Week 52 to Week 304
  To assess impact of long-term treatment on B-cell depletion.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (179):
- United States (32):
  - Providence Medical Foundation, Fullerton, California
  - Advanced Medical Research, La Palma, California
  - Medvin Clinical Research, Van Nuys, California
  - Bay Area Arthritis And Osteoporosis, Brandon, Florida
  - GNP Research, Cooper City, Florida
  - Sarasota Arthritis Res Ctr, Sarasota, Florida
  - West Broward Rheumatology Associates Inc, Tamarac, Florida
  - Augusta University Georgia, Augusta, Georgia
  - North GA Rheumatology Group PC, Suwanee, Georgia
  - Clin Invest Specialists Inc, Orland Park, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Ochsner Health System, Baton Rouge, Louisiana
  - The John Hopkins Jerome L Greene Sjogren, Baltimore, Maryland
  - Tufts School of Dental Medicine, Boston, Massachusetts
  - Arthritis Osteoporosis Assoc of NM, Las Cruces, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - St Lawrence Health System, Potsdam, New York
  - On Site Clinical Solutions Llc, Charlotte, North Carolina
  - Arthritis and Osteoporosis, Charlotte, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - STAT Research Inc, Dayton, Ohio
  - RAO Research LLC, Oklahoma City, Oklahoma
  - Altoona Center for Clin Res, Duncansville, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Shelby Research LLC, Memphis, Tennessee
  - Precision Comprehensive Research, Colleyville, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Houston Rheumatology & Arthrit, Katy, Texas
  - First Outpatient Research Unit, San Antonio, Texas
  - Advanced Rheumatology of Houston, Spring, Texas
  - Arthritis Northwest PLLC, Spokane, Washington
- Argentina (5):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, San Miguel Tucuman, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
- Australia (3):
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Woodville South, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
- Novartis Investigative Site, Graz, Austria
- Novartis Investigative Site, Leuven, Belgium
- Brazil (6):
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Bulgaria (2):
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Sofia
- Canada (5):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Sydney, Nova Scotia
  - Novartis Investigative Site, Rimouski, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Chile (4):
  - Novartis Investigative Site, Concepción, Bio Bio
  - Novartis Investigative Site, Valdivia, Los Ríos Region
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
- China (20):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Pingxiang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Linyi, Shandong
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Yinchuan, The Ningxia Hui Autonomous Reg
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Xinxiang
- Colombia (4):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bucaramanga, Santander Department
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Uherské Hradiště
- France (8):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Priest-en-Jarez
- Germany (9):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Ludwigshafen
- Novartis Investigative Site, Athens, Greece
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City
  - Novartis Investigative Site, Quetzaltenango
- Hungary (5):
  - Novartis Investigative Site, Székesfehérvár, Fejér
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Szeged
- India (2):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, New Delhi
- Israel (2):
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
- Italy (4):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Napoli
- Japan (12):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kuwana, Mie-ken
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Meguro-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Novartis Investigative Site, Vilnius, Lithuania
- Mexico (5):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, México
- Poland (7):
  - Novartis Investigative Site, Poznan, Greater Poland Voivodeship
  - Novartis Investigative Site, Krakow, Lesser Poland Voivodeship
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (3):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Guarda
  - Novartis Investigative Site, Lisbon
- Romania (3):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (3):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Zvolen
- South Africa (2):
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, Stellenbosch, Western Cape
- South Korea (2):
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (10):
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Stockholm, SE, Sweden
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara, Bilkent Cankaya
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Kocaeli
- United Kingdom (5):
  - Novartis Investigative Site, Doncaster
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Swindon

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com